CLINICAL TRIAL: NCT04840368
Title: Cardiovascular Risk and Functional Responses From Dancing at Home Compared With Walking in Elderly Individuals With and Without Type 2 Diabetes Mellitus: A Randomized Controlled Trial.
Brief Title: Cardiovascular Risk and Functional Responses From Dancing at Home in the Elderly With and Without Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Alvaro Reischak-Oliveira, Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 27116919.5.0000.5347
Record Dates: First submitted 2021-03-25; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Aging; Type2 Diabetes
Keywords: Aging; Type 2 diabetes; Aerobic Exercise; Dance; Cardiovascular risk; Functionality
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dancing (Experimental): Participants randomized to the dance group will take part in a dance intervention programme for 12 weeks, including 3 sessions per week (non-consecutive days), each lasting 60 min. Dance classes will be performed individually at home, guided by an expertise instructor, as live sessions online. They will include a variety of rhythms such as salsa, merengue, jazz dance, aerobics, etc. The dance sessions will include a warm up of approximately 10 min (posture, join mobility and dance technique), a main part of 40 min (practicing isolated dance moves and learning of specific choreographic routines), and a cool down of 10 min (muscle stretching and relaxation).
  Interventions: Other: Dancing
- Walking (Active Comparator): Participants randomized to the walking group will take part in a walking intervention programme for 12 weeks, including 3 sessions per week (non-consecutive days), each lasting 60 min. The walking session will include a warm up of 10 min (posture and join mobility), a main part of 40 min, and a cool down of 10 min (muscle stretching and relaxation). They will be performed individually, outside, at a self-selected intensity, with no supervision.
  Interventions: Other: Dancing

INTERVENTIONS:
Other: Dancing — Participants randomized to the dance group will take part in a dance intervention programme for 12 weeks, including 3 sessions per week (non-consecutive days), each lasting 60 min. Dance classes will be performed individually at home, guided by an expertise instructor, as live sessions online. They will include a variety of rhythms such as salsa, merengue, jazz dance, aerobics, etc. The dance sessions will include a warm up of approximately 10 min (posture, join mobility and dance technique), a main part of 40 min (practicing isolated dance moves and learning of specific choreographic routines), and a cool down of 10 min (muscle stretching and relaxation).

SUMMARY:
The goal of this randomized controlled trial is to investigate the effects of a dance intervention performed at home, on cardiovascular risk factors and functional capacity of elderly individuals with and without type 2 diabetes mellitus. Comparison will be performed with a walking exercise intervention, performed outside. Dance sessions will be guided online by an expertise instructor, and walking sessions will be performed at a self-selected intensity, with no simultaneous supervision. All participants will complete an exercise diary after each exercise session (reporting perception of subjective effort, affective responses, and others).The participants will include men and women between 65 and 80 years old, with body mass index inferior to 35 Kg /m2. The main outcome of this study is the peak oxygen consumption (VO2peak). The secondary outcomes are cardiovascular risk associated factors (C-reactive protein, TNF-alpha, lipid profile, etc) and functional performance (muscle strength and power, balance, gate ability, etc). Cognitive skills (executive function and memory) will be also assessed. The experimental design will include a control period of four weeks, two sessions of assessments before and after the interventions, and twelve weeks of dancing or walking interventions, performed three times a week, in non-consecutive days, with 60 min duration.

DETAILED DESCRIPTION:
The aging process is characterized by a loss of lean mass simultaneously to an increase in visceral adipose tissue (Bruseghini P. et al. 2015). This may result in reduced glucose uptake and increased levels of pro inflammatory cytokines, which leads to a chronic low grade inflammation state, insulin resistance, type 2 diabetes mellitus (T2DM) and elevated cardiovascular risk (CVR) (Krause, M.S. et al. 2013). Reductions in lean mass are also associated with reductions in muscle strength and power, inducing functional declines that result in difficulties to perform daily activities, and eventual loss of physical independence (Cadore, E.L. and Izquierdo, M. 2013) Costs with the treatment of aging-associated comorbidities are elevated for the health systems (Bielemann, R.M.K. et al. 2010). Searching for low cost strategies of prevention, with long term results, is essential then, especially the ones which may prevent dependence in a large spectrum (at the physical, social and cognitive levels), such as dancing (Laddu, D.R. et al 2020). Particularly, due to the pandemic of Corona Virus Disease-19 (COVID-19), long periods of self-isolation and social distancing have resulted in dramatic changes in the lifestyle of this population, beyond the risk of viral infection (Laddu, D.R. et al 2020). In this context, regular physical activity is considered to be a preventive strategy against chronic diseases due to its beneficial effects on global health (physical, mental, and social domains) (Fletcher, G.F. et.al. 2018). Particularly, dancing has been suggested as a strategy to increase levels of physical activity during quarantine periods (Jiménez-Pavón, D. et al. 2020), considering they can be adjusted for different ages, physical limitations, and levels of previous experience (Rodrigues-Krause, J.C. et al. 2019).

Therefore, the goal of this randomized controlled trial is to investigate the effects of a dance intervention on cardiovascular risk factors and functional capacity of older people, with and without type 2 diabetes mellitus (T2DM), comparing dancing to an active control group of walking exercise. The participants will include men and women between 65 and 80 years old, with body mass index inferior to 35 Kg /m2 and independent for performing daily activities. They should not be engaged in any type of regular physical activity in the past 6 months. Exclusion criteria will include cardiovascular complications, mobility limitations and neurodegenerative diseases.

The experimental design will include 3 parts: 1) Pre-intervention assessments: medical evaluation, fasting blood exams, maximum exercise test, assessments of body composition, balance, gate ability, muscular strength and power. 2) Control Period: 4 weeks for the follow up of the maintenance or changes in the primary and secondary outcomes responses of the participants. Primary and secondary outcomes will be evaluated before and after the control period. 3) Period of interventions: patients will be randomized in blocks (randomization.com), in accordance to their VO2peak, gender, and the presence of T2DM, to one of the two groups: dance or walking. The duration of the dance and walking interventions will be 12 weeks, including 3 sessions per week, each lasting 60 min. performed at home, guided by an expertise instructor, as live online sessions. Session will include several styles (salsa, jazz, aerobics), basic technical elements, no partner required. Walking: performed as a continuous aerobic exercise, outside, at a self-selected intensity, with no simultaneous supervision. Both interventions will include a warm-up (10 min), main part (40 min) and cool-down (10 min). All participants will complete an exercise diary after each exercise session (reporting perception of subjective effort, affective responses, and others). 3) Post-intervention assessments: the same protocols of testing of the pre-interventions assessments will be repeated. 4) Follow-up assessments: participants will be evaluated in 12 weeks times, for primary and secondary outcomes, after the end of the exercise intervention period.

The main outcome of this study is the peak oxygen consumption (VO2peak), as it has been associated with both, cardiovascular risk and functional performance in aging individuals. The secondary outcomes are: (1) cardiovascular risk associated factors: C-reactive protein, TNF-alpha, triglycerides, total cholesterol, LDL-cholesterol, HDL-cholesterol, fasting glucose and insulin, and homeostatic model assessment of insulin resistance (HOMA-IR). (2) Functional performance: muscle strength and power, balance, gate ability and muscle quality. (3) Cognitive function: executive function (random number generation and trial making test). In the following outcomes description of this Clinical Trials record, protocols of assessment for outcomes 1 to 20 are based on Rodrigues-Krause, J.C. et al. 2018. For outcomes 21 and 22 the reference is Forte, R. et al. 2013.

Results will be expressed in mean and confidence interval. All the assessments will be held at the Laboratory of Research in Exercise (LAPEX-UFRGS). Statistics: Generalized estimating equations, followed by the post hoc of least significant difference (LSD) (p<0.05). Comparisons before and after the interventions will be made among groups 1=dancing, 2=dancing T2DM, 3=walking, 4=walking T2DM.

Considering the well known benefits of the exercise, it is expected that our interventions will result in improvements on CVR (increases in cardiorespiratory fitness, reductions in adiposity, lipemia, insulin resistance and systemic inflammation), functionality (muscle strength and power, balance, gate and flexibility), and cognitive function (executive function). Our results will add on knowledge regarding the magnitude of possible gains from dancing at home, when compared to other forms of traditional aerobic exercise, a lack in the literature so far. Finally, the application of a purpose for an intervention of low cost and high levels of adherence, which stimulates multiple factors that decline with aging, may be a step forward in terms of strategies of prevention of aging-associated diseases on the public health context.

ELIGIBILITY:
Inclusion Criteria:

* Women and Men between 65 and 80 years old
* BMI inferior to 35 kg/m2
* Independent for performing daily activities (OARS scale)
* Not engaged in any type of regular exercise programme for the past 6 months
* Participants with T2DM should be previously diagnosed, with basal glycaemia superior to 126 mg/dL, and/or HbA1C superior to 6.5%.

Exclusion Criteria:

* Chronic diseases such as fibromyalgia, labyrinthitis, cancer or neurodegenerative disorders
* Compromised cognitive skills: Mini Mental State Examination (MMSE) scores inferior to 24/30.
* Bone, joints or muscle problems that could impair exercise performance
* Not being able to perform the effort test in the first assessment session, abnormal electrocardiogram, or any other condition identified by the physician of the study that limit the engagement in an exercise training programme.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-05-03 (Estimated); Primary Completion 2023-05-03 (Estimated); Study Completion 2023-12-23 (Estimated)

PRIMARY OUTCOMES:
Changes in Peak Oxygen Consumption (VO2peak), expressed in mL/Kg/min | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  Participants' VO2peak will be determined through an incremental exercise test on a treadmill. The test will start with a 5 min warm-up (from 3 to 5 km/h, increasing 0.5 km/h each min, until 5 min), followed by 2% increases in slope every min, while maintaining a constant speed of 5 km/h throughout the entire test. In order to be considered a maximum effort test, participants must attain at least two of the following criteria: (1) age-predicted HRmax, (2) respiratory exchange ratio (RER) ≥1.1, (3) subjective perception of effort ≥17 (Borg scale 6-20), (4) signals of muscle fatigue, such as loss of motor coordination. Ventilatory parameters will be measured continuously, breath-by breath, using an open-circuit spirometry system (Quark Cardio Pulmonary Exercise Test, Cosmed Italy). VO2peak was identified as the highest VO2 value in a line of tendency plotted against the time. Higher VO2peak values indicate better cardiorespiratory fitness and cardiovascular health.

SECONDARY OUTCOMES:
Changes in Triglycerides, expressed in milligrams per deciliter (mg/dL) | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  Triglycerides, a lipid profile marker, will be analyzed in plasma (after 8h fasting), and measured by enzymatic colorimetric method, using an automated analyzer (Cobas C111, Roche Diagnostics, Basel, Switzerland). Lower triglycerides values correspond to better metabolic health, as follows: Desirable levels: less than 150 (mg/dL). Borderline high: 150 to 199 mg/dL. High: 200 to 499 mg/dL.
Changes in Total Cholesterol, expressed in mg/dL | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  Total cholesterol, a lipid profile marker, will be analyzed in plasma (after 8h fasting), and measured by enzymatic colorimetric method, using an automated analyzer (Cobas C111, Roche Diagnostics, Basel, Switzerland). Lower LDL-Cholesterol values correspond to better metabolic health, as follows: Desirable: less than 200 mg/dL. Borderline high: 200-239 mg/dL. High: 240 mg/dL and above.
Changes in Low Density Lipoprotein Cholesterol (LDL-Cholesterol), expressed in mg/dL | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  LDL-Cholesterol levels, a lipid profile marker, will be estimated by Friedewald (1972). Lower LDL-Cholesterol values correspond to better metabolic health, as follows: Desirable: less than 100 mg/dL. Near-desirable: 100-129 mg/dL. Borderline High: 130-159 mg/dL. High: 160-189 mg/dL.
Changes in High Density Lipoprotein Cholesterol (HDL-Cholesterol), expressed in mg/dL | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  HDL-Cholesterol, a lipid profile marker, will be analyzed in plasma (after 8h fasting), and measured by enzymatic colorimetric method, using an automated analyzer (Cobas C111, Roche Diagnostics, Basel, Switzerland). Higher HDL-Cholesterol values correspond to better metabolic health, as follows: Desirable HDL-Cholesterol values: 45 to 70 mg/dL for men, 50 to 90 mg/dL for women.
Changes in Fasting Glycemia, expressed in mg/dL | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  Blood fasting glucose levels, a glycemic profile marker, will be analyzed in plasma (after 8h fasting), and measured by enzymatic colorimetric method, using an automated analyzer (Cobas C111, Roche Diagnostics, Basel, Switzerland). Normal values of fasting glycaemia is between 70 and 100 mg/dL for people who do not have diabetes. Fasting blood glucose levels greater than or equal to 126 mg/dL is considered for diagnosis of diabetes.
Changes in Fasting Insulin, expressed in milli-international units per litre (mlU/L) | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  Fasting insulin, a glycemic profile marker, will be analyzed in plasma (after 8h fasting), and determined by enzyme-linked immunosorbent assay (ELISA), according to manufacturer's instructions. Normal insulin levels are considered superior to 25 mlU/L, or < 174 pmol/L (SI Units: Conversional units x 6.945).
Changes in HOMA-IR, expressed in u.a | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  Glycemic profile marker. Homeostatic model of insulin resistance, calculated using fasting values of insulin and glycemia, in accordance with the following formula: fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.
Changes in Glycemic Responses to Oral Glucose Tolerance Test, expressed in mg/dL | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  Changes in Glycemic Responses to Oral Glucose Tolerance Test, used to test glucose tolerance, will be analyzed in plasma (after 8h fasting), by enzymatic colorimetric method, using an automatic analyzer (ROCHE, Cobas C111, Switzerland). Blood glucose will be measured at fasting, 30 min, one hour and two hours, after the ingestion of a drink with 75g of glucose dissolved in water. After two hours, plasma glucose levels (mg/dL) of 139 and below are considered normal. Values in between 140 and 199 correspond to pre-diabetes (impaired glucose tolerance). Values of 200 and above correspond to diabetes mellitus.
Changes in C-reactive protein (CRP), expressed in mg/L | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  CRP, a cardiovascular risk and inflammatory marker, will be analyzed in plasma (after 8h fasting), and determined by enzyme-linked immunosorbent assay (ELISA), according to manufacturer's instructions. High levels of CRP occur when some type of inflammatory or infectious processes is occurring in the bod. High CRP levels may predict a higher risk for cardiovascular disease. Values in between 3.0 to 10.0 mg/L indicate slight inflammation, but origin is unspecific.
Changes in Tumor necrosis factor alpha (TNF-alpha), expressed in pg/mL | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  TNF-alpha, an inflammatory marker, will be analyzed in serum (after 8h fasting), and determined by enzyme-linked immunosorbent assay (ELISA), according to manufacturer's instructions. Chronically elevated levels of TNF-alpha are linked with an increased risk of autoimmune diseases, obesity, and diabetes, among other diseases characterized by a chronic low-grade inflammation state. The recommended reference range of serum TNF-α vary from non detectable to 8.1 pg/mL.
Changes in Muscle Strength, expressed in (N・m) | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  The maximal isometric and isokinetic knee extension capacity will be measured using an Isokinetic Dynamometer (Cybex Norm, Cybex Norm,Ronkonkoma, New York, USA). The participants will perform 3 sets of 5 s and will be instructed to isometrically produce the maximal knee extension force as fast as possible at 60° of knee flexion (0° represents full extension). After a pre-test of 3 submaximal repetitions for angular velocity familiarization, maximal isokinetic knee extension peak torque will be measured during one set of 4 repetitions at the angular velocity of 60・s-1. The test will be performed in a 90° range of motion Both maximal isometric and isokinetic sets will be performed with 3 min of rest between them.
Changes in Muscle Power, expressed by the height (in cm) of the counter movement jump (CMJ) | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  Participants will perform a jump test using an electronic contact mat system. Jump height will be determined using an acknowledged flight-time calculation. Each participant will be instructed to use maximum effort to perform the double-leg CMJ test. They will be given 3 attempts to obtain their maximum jump height in each test, with 10 s of rest between attempts, with the highest value utilized for subsequent analysis.
Changes in Muscle Thickness, expressed in mm | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  For muscle thickness, transversal images of the right vastus lateralis, rectus femoris, vastus intermedius, and vastus medialis muscles will be obtained using a 38-mm, 9.0 megahertz linear-array transducer, with a Nemio XG ultrasound (Toshiba, Japan). The ultrasound muscular images were analysed via ImageJ software (National Institute of Health, USA, version 1.37). The subcutaneous adipose tissue and bone tissue will be identified, and the distance between them will be defined as muscle thickness. Quadriceps femoris muscle thickness will be considered as the sum of the four lower-body muscles muscle thickness. Increases in muscle thickness indicate gains in lean mass, improved body composition, and health and function related factors.
Changes in Static Balance, expressed by the time (in seconds) spent at an unipedal stance leg position | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  Static balance will be evaluated with the participant in unipedal stance of the dominant leg, with eyes closed. The opposite leg remained in the air, with hip and knee flexed at a 90° angle. The longest duration keeping the position (30s maximum) in three attempts will be recorded (stopwatch), with 2 min break.
Changes in Gait ability, measured by the Time to Up and Go (TUG) test | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  The TUG test consist in measuring the time (s) that the participant need to get up from a standard arm chair (43 cm), walk for 3m at usual walking speed, turn, and walk back to sit down. The fastest time in three attempts was recorded, with 2 min break in between them. Times were recorded to the nearest millisecond and transformed in m/s. A TUG score of 13.5 seconds or longer is predictive of reduced dynamic balance and fall risk.
Changes in Sit and Stand ability, expressed in seconds | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  The ability to seat and stand (chair raise test) will be assessed by the time required to rise from sitting five times as fast as possible from a standard chair (43 cm) with the participants folding arms across their chest. Recordings will be made using a stopwatch starting at the initiation of the movement and stopping when subjects stood upright for the 5th time.
Changes in the Fear of Falling, analyzed by the Falls Efficacy Scale- International Brazil (FES-I-Brazil). | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  The fear of falling will be analyzed by the Falls Efficacy Scale- International Brazil (FES-I-Brazil). This scale evaluates how confident the participant is in performing daily activities. The total score varies from 16 points (not worried at all) to 64 (extremely worried). The cut-off point to discriminate fallers and non fallers is 31 points.
Changes in Quality of Life, assessed by how the person feels in the physical, psychological, social and environmental domains of the World Health Organization Quality of Life (WHOQOL) questionnaire | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  Quality of life will be assessed by the abbreviated version of the World Health Organization Quality of Life (WHOQOL) questionnaire, which is specific for the elderly population. It contains 26 questions in total (2 for general quality of life assessment), and 24 including four domains (physical, psychological, social and environmental). The scores for each question are from 1 (very bad) to 5 (very good) quality of life for each specific domain. Scores 2, 3 and 4 mean bad, neutral and good, respectively. The final score is expressed in percentage (from 0 to 100%). As closer the score is to 100%, higher is the general quality of life of that individual.
Changes in Leisure Time Physical Activity | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  The Godin-Shephard leisure-time physical activity questionnaire will be used in its validated version and translated into Brazilian Portuguese. Light, moderate or vigorous physical activities, performed for at least 15 min during leisure time, will be registered by the participants. The frequency is multiplied by the metabolic equivalent (MET). High scores indicate a higher level of physical activity during leisure. For example, in the reference to the score in units using only moderate and strenuous physical activities, 24 units or more means "Active", indicating substantial benefits; from 14 to 23 units means "Moderately active", indicating some benefits; and less than 14 units means "Insufficiently active", indicating low benefits.
Change in Executive function, assessed by the Random number generation task | before intervention (week 0), after control period (week 5), and after intervention (week 13)
  The random number generation task evaluates executive functions, particularly inhibition. Briefly, participants verbally generated a random sequence of 100 numbers chosen between one and nine, at a frequency of 40 bpm, paced by a metronome. The randomness of the sequence is elaborated to obtain three indices that were theoreti¬cally related to the inhibitory function: the Turning Point Index, the Adjacency, and the Runs. High levels on the Turning Point Index, but low levels of Adjacency and Runs correspond to a high ability to inhibit the production of stereotyped strings, therefore contributing to the optimal control of complex activities.
Change in Executive function, assessed by the Trail making test | [Time Frame: before intervention (week 0), after control period (week 5), and after intervention (week 13)]
  The trail making test assesses attention, speed, and cognitive flexibility. The standard protocol used requires participants to draw lines connecting in ascending order and as quickly as possible 25 circles distributed over a sheet of paper. The test has a part A with numbers only and a part B with numbers and letters joined in alternation (i.e, 1-A-2-B-3-C, and so on). A summary score will be calculated by subtracting the time taken in seconds to complete part A from the time at part B (ΔTrail Making) and used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Reischak-Oliveira, PhD, Principal Investigator — Federal University of Rio Grande do Sul; Josianne Rodrigues-Krause, PhD, Study Director — Federal University of Rio Grande do Sul
Locations (1):
- School of Physical Education, Physiotherapy and Dance (Universidade Feferal do Rio Grande do Sul), Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Yes
We intend that the data to be collected in this trial may contribute beyond our actions to the knowledge on dance, exercise, aging and T2DM. Ethical consent from participants, and Institutional Review Boards approval to share data will be obtained. Data sets, variables' dictionary and statistical analysis description will be available online upon registration and acceptance of the study team's data sharing terms and policy. Data usage will be under the PI's auspices, but restrictions or screenings will not be imposed upon data requests. VO2peak (main outcome) data and relevant support information (sociodemographic, clinical history and allocated groups) will be shared. Data on other outcomes may be requested by contacting the PI.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be shared through a public repository no later than six months after the first study publication (data access available as long as deemed necessary by the study coordination).
Access Criteria: The public repository for data sharing is not yet defined (it will be presented in the study website and scientific publications).

REFERENCES:
- [Background] Bruseghini P, Calabria E, Tam E, Milanese C, Oliboni E, Pezzato A, Pogliaghi S, Salvagno GL, Schena F, Mucelli RP, Capelli C. Effects of eight weeks of aerobic interval training and of isoinertial resistance training on risk factors of cardiometabolic diseases and exercise capacity in healthy elderly subjects. Oncotarget. 2015 Jul 10;6(19):16998-7015. doi: 10.18632/oncotarget.4031. PMID 26046575
- [Background] Krause M, Rodrigues-Krause J, O'Hagan C, Medlow P, Davison G, Susta D, Boreham C, Newsholme P, O'Donnell M, Murphy C, De Vito G. The effects of aerobic exercise training at two different intensities in obesity and type 2 diabetes: implications for oxidative stress, low-grade inflammation and nitric oxide production. Eur J Appl Physiol. 2014 Feb;114(2):251-60. doi: 10.1007/s00421-013-2769-6. PMID 24233244
- [Background] Cadore EL, Izquierdo M. How to simultaneously optimize muscle strength, power, functional capacity, and cardiovascular gains in the elderly: an update. Age (Dordr). 2013 Dec;35(6):2329-44. doi: 10.1007/s11357-012-9503-x. Epub 2013 Jan 4. PMID 23288690
- [Background] Bielemann, R.M.K., A. G; Hallal, P.C. R, Physical activity and cost savings for chronic diseases to the sistema Único de saúde. Revista Brasileira de Atividade Física e Saúde, 2010. 15(1): p. 9-14.
- [Background] Laddu DR, Lavie CJ, Phillips SA, Arena R. Physical activity for immunity protection: Inoculating populations with healthy living medicine in preparation for the next pandemic. Prog Cardiovasc Dis. 2021 Jan-Feb;64:102-104. doi: 10.1016/j.pcad.2020.04.006. Epub 2020 Apr 9. No abstract available. PMID 32278694
- [Background] Fletcher GF, Landolfo C, Niebauer J, Ozemek C, Arena R, Lavie CJ. Promoting Physical Activity and Exercise: JACC Health Promotion Series. J Am Coll Cardiol. 2018 Oct 2;72(14):1622-1639. doi: 10.1016/j.jacc.2018.08.2141. PMID 30261965
- [Background] Jimenez-Pavon D, Carbonell-Baeza A, Lavie CJ. Physical exercise as therapy to fight against the mental and physical consequences of COVID-19 quarantine: Special focus in older people. Prog Cardiovasc Dis. 2020 May-Jun;63(3):386-388. doi: 10.1016/j.pcad.2020.03.009. Epub 2020 Mar 24. No abstract available. PMID 32220590
- [Background] Rodrigues-Krause J, Krause M, Reischak-Oliveira A. Dancing for Healthy Aging: Functional and Metabolic Perspectives. Altern Ther Health Med. 2019 Jan;25(1):44-63. PMID 29428927
- [Background] Rodrigues-Krause J, Farinha JB, Ramis TR, Macedo RCO, Boeno FP, Dos Santos GC, Vargas J Jr, Lopez P, Grazioli R, Costa RR, Pinto RS, Krause M, Reischak-Oliveira A. Effects of dancing compared to walking on cardiovascular risk and functional capacity of older women: A randomized controlled trial. Exp Gerontol. 2018 Dec;114:67-77. doi: 10.1016/j.exger.2018.10.015. Epub 2018 Oct 31. PMID 30389581
- [Background] Forte R, Boreham CA, Leite JC, De Vito G, Brennan L, Gibney ER, Pesce C. Enhancing cognitive functioning in the elderly: multicomponent vs resistance training. Clin Interv Aging. 2013;8:19-27. doi: 10.2147/CIA.S36514. Epub 2013 Jan 10. PMID 23341738